CLINICAL TRIAL: NCT07387315
Title: A Randomized, Placebo Controlled Trial of Nitrous Oxide/Oxygen Plus Standard Care Versus Standard Care Alone During In-office Intradetrusor onabotulinumtoxinA (Botox) Injections
Brief Title: A Randomized, Placebo-controlled Trial of Nitrous Oxide During In-office Bladder Botox Injections
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-130
Record Dates: First submitted 2026-01-28; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Overactive Bladder; Neurogenic Bladder; Urge Incontinence; Pain; Urinary Incontinence; Urinary Bladder, Overactive; Urinary Bladder, Neurogenic; Urinary Bladder Neurogenesis; Urinary Incontinence, Urge; Pelvic Floor Disorders
Keywords: Overactive Bladder; Urinary Incontinence; Urge Incontinence; Intradetrusor Injection; OnabotulinumtoxinA; Botox; Bladder Botox; Botulinum Toxins, Type A; Pain Management; Analgesia; Nitrous Oxide; Office-based Procedures; Urogynecology; Pelvic Floor Disorder
MeSH Terms: conditions — Urinary Bladder, Overactive; Urinary Bladder, Neurogenic; Urinary Incontinence, Urge; Pain; Urinary Incontinence; Pelvic Floor Disorders; Agnosia | interventions — Nitrous Oxide; Oxygen; Standard of Care; Lidocaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be masked to sham mask versus mask with nitrous oxide/oxygen. Masking of the investigators would not be feasible given the use of participant self-administered inhaled nitrous oxide gas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham Mask Plus Standard Care (Active Comparator): The sham mask plus standard care group will receive a mask that is connected to the Pro-Nox system but with the valves turned completely off; therefore they will inhale room air plus standard care: intravesical instillation of 1-2% lidocaine solution (30-50 mL) with at least 15 minutes dwell time before the procedure.
  Interventions: Drug: Standard Care for Bladder Botox Injection; Other: Sham Mask
- Nitrous Oxide Plus Standard Care (Experimental): Participants in this group will receive standard care plus 50:50 mix of inhaled nitrous oxide/oxygen self-administered using the Pro-Nox system during the bladder Botox procedure.
  Interventions: Drug: Pro-Nox Nitrous Oxide/Oxygen Delivery System; Drug: Standard Care for Bladder Botox Injection

INTERVENTIONS:
Drug: Pro-Nox Nitrous Oxide/Oxygen Delivery System — The Pro-Nox system delivers a fixed 50:50 mixture of nitrous oxide and oxygen for patient self-administered inhaled analgesia. Participants will self-administer nitrous oxide throughout the in-office bladder Botox procedure.
  Other Names: Pro-Nox; Nitrous oxide/oxygen 50:50 mixture; Nitrous oxide/oxygen; Nitrous; Nitrous oxide; Nitrous oxide analgesia
  Arms: Nitrous Oxide Plus Standard Care
Drug: Standard Care for Bladder Botox Injection — Standard care includes intravesical instilled 1-2% lidocaine with a dwell time of at least 15 minutes before the procedure.
  Other Names: Intravesical lidocaine; Lidocaine; Standard care; Standard analgesia; Local analgesia
Other: Sham Mask — The Sham Mask will involve that participant using the same mask as that of the Nitrous Oxide group, but connected to a Pro-Nox system that is turned completely off. They will therefore receive room air through the mask.
  Other Names: Placebo; Room Air
  Arms: Sham Mask Plus Standard Care

SUMMARY:
The goal of this clinical trial is to assess if a mix of nitrous oxide and oxygen can improve pain control during bladder Botox injections. The primary question it aims to answer is: Does using nitrous oxide lower the overall level of pain during the procedure?

Researchers will compare a 50:50 nitrous oxide/oxygen mixture (administered with the Pro-Nox system) plus standard care (with lidocaine in the bladder) to sham mask plus standard care to see if nitrous oxide works better for lowering pain.

Participants will:

* Receive their bladder Botox injection in the office setting
* Either use nitrous oxide/oxygen plus standard care during the procedure, or sham mask plus standard care
* Answer brief questions about pain, anxiety, satisfaction, and willingness to repeat the procedure

DETAILED DESCRIPTION:
This study will assess if a 50:50 nitrous oxide and oxygen mixture can lower pain in women undergoing in-office bladder onabotulinumtoxinA (Botox) injections. Many people report pain during this procedure, and pain is a common reason not to repeat the procedure. Nitrous oxide is a fast-acting inhaled analgesic that is used commonly in the office setting.

This randomized controlled trial will compare nitrous oxide/oxygen plus standard care with sham mask plus standard care. Participants assigned to the nitrous oxide group will receive nitrous oxide via the Pro-Nox device during the procedure. Both, participants assigned to the nitrous oxide group and the standard care alone group, will receive the usual lidocaine instilled in the bladder for at least 15 minutes.

The study will measure participants overall pain during the procedure. It will also assess peak pain, overall anxiety, satisfaction, willingness to repeat, interest in using nitrous oxide in future bladder Botox procedures, and side effects. Nitrous oxide is expected to wear off within minutes, allowing participants to leave the clinic without restrictions.

This research study would be first randomized-controlled trial to evaluate nitrous oxide for pain management during this common in-office procedure.

ELIGIBILITY:
Inclusion Criteria:

* Adult women ≥18 years old scheduled for in-office intradetrusor botulinum toxin injection and able to consent.

Exclusion Criteria:

* Known/suspected vitamin B12 or folate deficiency or high-risk state (e.g., pernicious anemia, malabsorption, post-bariatric or strict vegan without supplementation)
* currently pregnant
* severe/unstable pulmonary disease or baseline hypoxemia requiring supplemental home oxygen
* eye or ear surgery in the last six weeks
* trapped-air conditions (e.g., untreated pneumothorax, bowel obstruction)
* severe active otitis/sinus disease
* inability to follow directions
* history of adverse reaction to nitrous oxide

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Overall Pain (10-point NRS) | At least 3 minutes after completion of the procedure.
  Patient self-reported overall pain during the procedure on an 11-point numeric rating scale.

SECONDARY OUTCOMES:
Peak Pain (10-point NRS) | At least 3 minutes after completion of the procedure.
  Patient self-reported peak pain during the procedure on an 11-point numeric rating scale.
Peak Pain Timing | At least 3 minutes after completion of the procedure.
  Patient self-reported timing of peak pain during the procedure, as it corresponds to different steps during the procedure.
Overall Anxiety (10-point NRS) | At least 3 minutes after completion of the procedure.
  Patient self-reported overall anxiety during the procedure on an 11-point numeric rating scale.
Satisfaction with Pain Management (10-point NRS) | At least 3 minutes after completion of the procedure.
  Patient self-reported satisfaction with pain management during the procedure on an 11-point numeric rating scale.
Willingness to Repeat (5-point Likert) | At least 3 minutes after completion of the procedure.
  Patient self-reported willingness to repeat under similar pain and anxiety management conditions, on a 5-point Likert scale.

OTHER OUTCOMES:
Nitrous Interest (5-point Likert) | At least 3 minutes after completion of the procedure.
  Patient self-reported interest in use of nitrous oxide for pain and anxiety management in a future procedure, on a 5-point Likert scale.
Adverse Effects | Immediately following the procedure. Completed by performing surgeon.
  Physician reported adverse events encountered peri-operatively.
Blinding Assessment | At least 3 minutes after completion of the procedure.
  Patient self-reported perceived treatment assignment (nitrous oxide/oxygen vs sham mask), recorded as nitrous oxide, sham mask, or unsure.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Cincinnati Urogynecology Associates, Cincinnati, Ohio
  - Trihealth (Good Samaritan Hospital, Bethesda North Hospital), Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
Do not plan to share individual participant data with other researchers.